CLINICAL TRIAL: NCT07324928
Title: Evaluate and Compare the Effect of Ferric Sulphate and Putty MTA as Pulpotomy Agent in Vital Primary Teeth
Brief Title: Effect of Ferric Sulphate and Putty MTA as Pulpotomy Agent in Vital Primary Teeth
Acronym: CT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, satish vishwanathaiah, Associate professor, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Jazan college of Dentistry
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Pulptomy; Dental Caries; Pulp Therapy
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Ferric Sulphate) (Experimental): already described
  Interventions: Procedure: Ferric sulphate
- Group B ( Putty MTA) (Experimental): already described
  Interventions: Procedure: Putty MTA

INTERVENTIONS:
Procedure: Ferric sulphate — already described
  Arms: Group A (Ferric Sulphate)
Procedure: Putty MTA — already described
  Arms: Group B ( Putty MTA)

SUMMARY:
The pulp in primary teeth has a high potential for repair because of high degree of cellularity and vascularity. The rationale for the pulpotomy procedure is that the radicular pulp tissue is healthy and capable of healing after surgical amputation of the affected or the infected coronal pulp. There is ample information about pulpotomy in deciduous molars using formocresol, glutaraldehyde, electrosurgery, ferric sulphate, calcium hydroxide, MTA etc. The vital pulpotomy process using formocresol has been widely accepted in primary tooth pulp therapy because of its simplicity and good prognosis. However, much concern as arisen over the mutagenic and carcinogenic potential of formaldehyde containing products, the cytotoxic effects of formocresol and the possible diffusion into the surrounding and systemic tissues. In order to avoid the possible harmful effects of formocresol; other pulpotomy agents for vital pulpotomy procedure is being sought such as ferric sulphate and MTA with promising results due to their advantages such as devitalization and regenerative agents respectively.

Ferric sulphate [Fe2(SO4)3] as a 15.5% solution is a coagulative and local hemostatic agent.

Ferric sulphate is a material with minimal devitalization and non-induction of pulp tissue. It is used as a coagulative and hemostatic retraction agent. Ferric sulfate is proposed as a pulpotomy agent on the theory that its mechanism of controlling hemorrhage might minimize the chances for inflammation. Ranly proposes the possibility that the metal-protein clot at the surface of the pulp stumps may act as a barrier to the irritative components of the sub-base which helps in minimizing the complications from the material. The hemostatic properties of ferric sulfate and the favorable pulpal response make it a promising medicament for pulpotomy. Erdem AP et al in their study observed no significant differences among 3 experimental materials MTA, Formocresol and Ferric sulphate. Fei AL et al observed clinical ad radiographic success than the Formocresol group at the end of one year.

Mineral trioxide aggregate (MTA) is one such regenerative material recognized as the reference material for conservative pulp vitality treatments in primary teeth, with high pulpotomy success rates (90%-100%) in clinical, radiographic, and histopathologic studies. However, MTA has difficult handling characteristics, contains heavy metals such as alumina and bismuth oxide, and is expensive. Technological improvements in the medical meteorology led to development and innovations in bioceramic nanotechnology (Bioceramics) which exhibit excellent biocompatibility with properties in unison with hydroxyapatite. Recently, bioceramic putty, a calcium silicate based nanoparticulate material, was introduced into dentistry as a root repairing material. It is an insoluble, radiopaque, aluminum free, and zirconium oxide incorporated material developed for potential dental surgery applications. Moreover, it stimulates the deposition of hydroxyapatite on its surface when exposed to tissue fluids, forms well organized dentin, and has low cytotoxicity. Despite its ease of handling, high viscosity, shorter setting time, better physical properties over MTA and the biomimetic property of bioceramics, its clinical application in the field of vital pulp therapy in primary teeth has not been explored so far. Kumar KR et al in their study showed clinical success rate of 95 % and radiographic success rate of around 90% with MTA.

Some studies have reported internal resorption seen with ferric sulphate pulpotomy, sensitivity, premature tooth loss , furcation radiolucency, gingival swelling but not attributed the exact reason for the same. They attributed to tooth selection for the procedure. Hence proper tooth selection is a criteria for the success of pulpotomy.

DETAILED DESCRIPTION:
Pilot study will not be conducted as we are not testing the feasibility of the methodology.

This study will be performed on 60 patients aged 6 to 10 years attending the clinics of department of paediatric dentistry, college of dentistry, Jazan university will be considered for the study.

Before starting; the procedure will be explained; verbal and written consent will be obtained by the parent or guardian. After obtaining consent a total of 60 molars will be randomly divided into two groups, Group A with ferric sulphate and Group B with Putty MTA using a lottery randomization technique.

Pulpotomy will be done in both the groups followed by GIC restoration. Immediate post operative radiograph will be taken for all the patients. The patients will be recalled at 1month and 3 month and 6-month interval for clinical and radiographic evaluation.

In recall visits all the teeth will be evaluated to grade them as either success or failure based on the clinical and radiographic criteria. This will be evaluated by investigators unaware of the group assignment.

Criteria for evaluating the success:

Teeth which presented with no symptoms of pain. Tenderness to percussion, swelling, fistulation, or pathologic mobility clinically as well as no evidence of radicular radiolucency, internal or external root resorption or periodontal ligament space widening radiographically will be considered successful. Any tooth which showed signs of symptoms of failure will be treated with pulpectomy

ELIGIBILITY:
Inclusion criteria

1. Healthy children with no systemic illness, allergies
2. Co-operative child
3. Patient requiring pulpotomy on deciduous molars with carious /mechanical pulp exposure
4. children with proper parental consent
5. No clinical or radiographical signs of pulp pathoses
6. Possibility of proper restoration of tooth after the procedure
7. Haemostasis should be easily achievable after pulp amputation

Exclusion criteria

1. Children with systemic illness and allergy
2. Un co-operative child
3. clinical or radiographical signs of pulp pathoses
4. unrestorable tooth
5. Haemostasis not achieved after pulp amputation

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Clinical criteria | 1 month, 3 month , 6 month
  Clinical Teeth which presented with
  * no symptoms of pain.
  * Tenderness to percussion,
  * swelling,
  * fistulation, or
  * pathologic mobility
Radiographic criteria | 1 month, 3 month, 6 month
  * Evidence of radicular radiolucency,
  * Internal or external root resorption
  * Periodontal ligament space widening

IPD SHARING:
Plan to Share IPD: No